CLINICAL TRIAL: NCT06913855
Title: The Effects of EMLA Cream and Cold Application on Pain, Fear and Vital Signs Before Chest Tube Removal in Children: a Randomized Controlled Trial
Brief Title: The Effects of EMLA Cream and Cold Application on Pain, Fear and Vital Signs Before Chest Tube Removal in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-61
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chest Tube Removal; Children; Pain Management
Keywords: Chest tube removal; Children; Pain management
MeSH Terms: conditions — Agnosia | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental and control groups using block randomization method. Age, sex and procedural fear variables will be used for block randomization. In order to reach the sample size calculated in the study, strata will be repeated two times (2X2X3X2) and 24 children will be included in each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, participants will be divided into 3 groups. A web-based randomization list creation tool will be used to create the blocked randomization list. Control and intervention groups will be coded as A, B and C using the sealed envelope method. Randomization information will be kept from the researcher involved in data collection until data collection begins. The researcher will learn which group each child is in just before the application (researcher blinding).
  Research data will be entered into the computer database by coding the group name as A, B and C, and statistical analysis will be performed using this coding (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): The chest tube removal procedure will be performed according to clinical routine practice.
- EMLA cream (Experimental): EMLA cream will be applied to the chest tube area 3 hours before the chest tube removal procedure. Then, the chest tube removal procedure will be performed.
  Interventions: Drug: EMLA Cream
- Cold application (Experimental): Before the chest tube removal procedure, an ice cube pack will be applied to the chest tube area. Cold application will continue until the skin temperature drops to 13.0 degrees. Then the chest tube removal procedure will be performed.
  Interventions: Procedure: Cold application

INTERVENTIONS:
Drug: EMLA Cream — EMLA cream is applied once, 3 hours before the tube is removed. EMLA cream will be applied by the researcher in a thin layer to an area of 7-10 cm2, with the chest tube entrance to the skin remaining in the center. It will be covered with a Tegaderm transparent film dressing.
  Arms: EMLA cream
Procedure: Cold application — Cold application will be made with an ice cube pack immediately before the chest tube removal procedure. Cold application will be applied to a 7 cm diameter area, with the chest tube entrance to the skin being considered as the center. Skin temperature will be measured with an infrared thermometer and will be ensured to reach 13.0 degrees. Ice pack application is expected to last approximately 9-10 minutes.
  Arms: Cold application

SUMMARY:
This study is being conducted to determine the effect of EMLA cream and cold application on pain, fear and vital signs before chest tube removal in children aged 7-18 years.

DETAILED DESCRIPTION:
A chest tube is a device used to drain air or fluid from the pleural cavity under sterile conditions by inserting a thin or thick tube. Chest tubes adhere to the endothelium of the chest cavity after insertion and while in place. For this reason, the pulling force applied when they are removed breaks these adhesions and causes intense, localised and transient acute pain. Chest tube removal pain, defined as one of the patient's worst life experiences related to the surgical procedure, is an iatrogenic pain caused by an invasive procedure. Therefore, chest tube removal is a painful, anxious and frightening experience for the patient. There are few studies of pharmacological and non-pharmacological methods of pain control during chest tube removal in children. However, the management of pain associated with surgical procedures in childhood is very important for the management of pain, anxiety and fear that children will experience with future medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Having two chest tubes (mediastinal/pleural) placed after open heart surgery
* Turkish literate
* With stable vital signs
* Willing to participate in the research

Exclusion Criteria:

* Experience with chest tube removal procedure
* Using analgesics other than routine procedures before the procedure
* Children receiving mechanical ventilation support
* Children who have complications in the postoperative period (heart and respiratory failure, repeated surgery, etc.)
* Children with a mental disability, perception problem, visual and hearing impairment
* Children with communication problems. • Children with cold allergies

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Procedural pain score- Wong-Baker FACES Pain Rating Scale | 3 hours before the procedure, immediately before the procedure, 1 minute after the procedure and 5 minutes after the procedure
  The scale is used to diagnose pain in children aged 3-18 years. It consists of six facial expressions, each one representing an increasing degree of pain scored on a scale 0 to 5 from left to right. The first face is a happy face representing "no pain=0" while the last face is a crying face representing "the worst pain imaginable=5". Higher scores indicate low pain tolerance. Participants are asked to choose the facial expression that best represents their pain.

SECONDARY OUTCOMES:
Procedural fear score- Children's Fear Scale (CFS) | 3 hours before the procedure, immediately before the procedure, 1 minute after the procedure and 5 minutes after the procedure
  The CFS was developed to measure fear and anxiety in children. It consists of five facial expressions that represent a range from neutral to extreme fear. It is scored between 0 and 4. Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedure.
Oxygen saturation | 3 hours before the procedure, immediately before the procedure, 1 minute after the procedure and 5 minutes after the procedure
  Children will be connected to a pulse oximeter monitor; oxygen saturation will be monitored before, during and after the procedure.
Pulse rate | 3 hours before the procedure, immediately before the procedure, 1 minute after the procedure and 5 minutes after the procedure
  Children will be connected to a pulse oximeter monitor; their pulse rate will be monitored before, during and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: July through December of 2026
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Rosen DA, Morris JL, Rosen KR, Valenzuela RC, Vidulich MG, Steelman RJ, Gustafson RA. Analgesia for pediatric thoracostomy tube removal. Anesth Analg. 2000 May;90(5):1025-8. doi: 10.1097/00000539-200005000-00005. PMID 10781447
- [Background] Pouraboli B, Mirlashari J, Fakhr AS, Ranjbar H, Ashtari S. The Effect of Facilitated Tucking on the Pain Intensity Induced by Chest Tube Removal in Infants. Adv Neonatal Care. 2022 Oct 1;22(5):467-472. doi: 10.1097/ANC.0000000000000936. Epub 2021 Aug 11. PMID 34387216